CLINICAL TRIAL: NCT03823339
Title: A Multicenter Prospective Non-interventional Study Investigating the Treatment Effect of Xultophy® Intensification in a Real World Population With Type 2 Diabetes in United Arab Emirates
Brief Title: A Research Study, Looking at How Xultophy® Works in People With Type 2 Diabetes in Local Clinical Practice in United Arab Emirates
Acronym: INTENSIFY
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9068-4458; U1111-1213-4338 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-01-24; First posted 2019-01-30 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with type 2 diabetes (T2DM): Patients with T2DM treated with any basal insulin or glucagon-Like peptide-1 receptor agonist (GLP-1 RA) (including once weekly GLP-1 RA) with/without oral antidiabetic drug (OAD) treatment, and with inadequate glycaemic control, for whom the physician had decided to intensify their treatment with Xultophy®
  Interventions: Drug: Insulin degludec/liraglutide

INTERVENTIONS:
Drug: Insulin degludec/liraglutide — Patients will be treated with Insulin degludec/liraglutide (Xultophy®) at the treating physician's discretion and independent from the decision to include the patient in the study.

SUMMARY:
The purpose of the study is to collect information on how Xultophy® works in patients with type 2 diabetes. The participants will get Xultophy® as prescribed to them by the study doctor. The study will last for about 26-34 weeks. The participants will be asked questions about their health and their diabetes treatment as part of their normal study doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available Xultophy® has been made by the patient/Legally Acceptable Representative and the treating physician before and independently from the decision to include the patient in this study.
* Male or female, age greater than or equal to 18 years at the time of signing informed consent.
* Diagnosed with type 2 diabetes and treated with basal insulin plus or minus oral anti-diabetic drugs (OADs) or Glucagon-Like Peptide-1 Receptor Agonist (GLP-1 RA) plus or minus OADs, except Xultophy®, for at least 12 weeks prior to informed consent and initiation visit (visit 1).
* Available and documented glycosylated haemoglobin A1c (HbA1c) value less than or equal to 12 weeks prior to initiation of Xultophy® treatment.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients as specified in the Xultophy® local label.
* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Female who is known pregnant, breast-feeding or intends to become pregnant.
* Treated with Xultophy® previously.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Type 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Change in laboratory measured glycosylated haemoglobin A1c (HbA1c) | From baseline [≤12 weeks prior to treatment initiation [week 0]) to end of study (26-34 weeks)
  Measured in % point

SECONDARY OUTCOMES:
Patients reached HbA1c less than 7% at end of study (Yes/No ) | At the end of study visit (26-34 weeks)
  Number of patients who achieved/not achieved HbA1c at end of study: <7.0%
Change in laboratory measured fasting plasma glucose (FPG) | From baseline [≤12 weeks prior to treatment initiation [week 0]) to end of study (26-34 weeks)
  Measured in mg/dL
Average dose step of Xultophy® at end of the study | At the end of study (26-34 weeks)
  Measured in dose steps/day
Change of body weight | From baseline [≤12 weeks prior to treatment initiation [week 0]) to end of study (26-34 weeks)
  Measured in kg
Change in number of patient self-reported overall non-severe hypoglycaemic episodes based on recollection | Pre- to post- initiation of treatment with Xultophy®. Episodes occurring within 4 weeks prior to initiation of treatment with Xultophy® and to within 4 weeks prior to end of study (26-34 weeks)
  Number of episodes
Change in number of patient self-reported nocturnal non-severe hypoglycaemic episodes based on recollection | Pre- to post- initiation of treatment with Xultophy®. Episodes occurring within 4 weeks prior to initiation of treatment with Xultophy® and to within 4 weeks prior to end of study (26-34 weeks)
  Number of episodes
Change in number of patient self-reported severe hypoglycaemic episodes based on recollection (overall) | Pre- to post- initiation of treatment with Xultophy®. Episodes occurring within 26 weeks prior to initiation of treatment with Xultophy® and to within 26 weeks prior to end of study (26-34 weeks)
  Number of episodes
Reason(s) for discontinuing treatment with Xultophy® during the treatment period, if applicable | At the end of study (26-34 weeks)
  Pre-specified response option(s)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (3):
- United Arab Emirates (3):
  - Novo Nordisk Investigational Site, Abu Dhabi
  - Novo Nordisk Investigational Site, Ajman
  - Novo Nordisk Investigational Site, Dubai

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com